CLINICAL TRIAL: NCT04406103
Title: Your Answers When Needing Sleep in New Brunswick (YAWNS NB): A Randomized Controlled Trial Comparing Sleepwell, EMPOWER, and Treatment as Usual for Benzodiazepine Receptor Agonist Discontinuation in Older Adults (Protocol)
Brief Title: Protocol - Your Answers When Needing Sleep in New Brunswick
Acronym: YAWNS NB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Gardner (Other)
Collaborators: University of New Brunswick (Other); Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, David Gardner, Professor, Dalhousie University
Organization: Dalhousie University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5184
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Insomnia Chronic
Keywords: insomnia; benzodiazepines; deprescribing; cognitive-behavioural therapy for insomnia (CBTi)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleepwell (Experimental): Mailed information package includes 2 Sleepwell booklets (How to get your sleep back and How to stop sleeping pills)
  Interventions: Behavioral: Sleepwell
- Empower (Active Comparator): Mailed information package includes 2 Empower booklets (You may be at risk AND How to get a good night's sleep without sleeping pills)
  Interventions: Behavioral: Empower
- TAU (No Intervention): Treatment-as-usual group: no mailed intervention package.

INTERVENTIONS:
Behavioral: Sleepwell — Information intended to support capability, opportunity, and motivation for stopping sleeping pill use and using non-pharmacological approaches to managing insomnia.
  Arms: Sleepwell
Behavioral: Empower — Information intended to support capability, opportunity, and motivation for stopping sleeping pill use and using non-pharmacological approaches to managing insomnia.
  Arms: Empower

SUMMARY:
New Brunswick has an aging population with Canada's highest rate of sleeping pill use. The rate of long-term (chronic) use among NB seniors is 25%, well in excess of the Canadian average of 10%. The rate of use is higher in women and increases with age, as do risks for serious harms.

Sleeping pills risks are substantial and costly, especially to seniors. Research does not support their long-term use. Risk for falls causing injuries, including hip fractures, is a leading concern. They impair mental and physical functioning resulting in a loss of independence and cause impaired driving and a higher rate of serious crashes. The rate of near-fatal and fatal overdoses from mixing sleeping pills with other drugs is on the rise. Stopping treatment can be difficult due to physical dependence and withdrawal symptoms.

Cognitive behavioural therapy for insomnia (CBTi) is recommended as the first-line treatment of chronic insomnia. Sleeping pills are only to be considered when CBTi fails. However, these recommendations are not reflected in primary care practice.

Internationally, many educational interventions targeting prescribers have been tried, yet have failed to reduce sleeping pill use. However, a 12-page pamphlet (EMPOWER) given directly to seniors in a clinical trial was associated with a large reduction in sleeping pill use. Using a similarly persuasive approach, Sleepwell (mysleepwell.ca) was developed to reduce the use of sleeping pills and facilitate CBTi access and use. Sleepwell differs from EMPOWER by providing specific information and recommendations regarding CBTi in addition to guidance on how to stop sleeping pills.

This study will evaluate the effectiveness of direct-to-patient interventions on long-term sleeping pill use.

DETAILED DESCRIPTION:
The investigators are proposing to investigate direct-to-patient health promotion interventions that promote sleeping pill dose reduction and treatment discontinuation by enhancing self-efficacy through various behaviour change techniques embedded in printed information provided to patients. Seniors will be invited to participate via direct telephone contact, information sharing through seniors' organizations, education sessions for seniors, and public notices. Prospective participants will be given the option of which way they would like to participate in the research:

Option 1: full participation including baseline interview, 6-month interview, and access to specific data from the participant's personal health record); Option 2: limited participation to baseline and 6-month interviews only; and Option 3: limited participation to baseline interview and access to specific data from the participant's personal health record.

This will form two sets of participants; those who do and those who do not permit access to outcomes from their personal health record. Participants that select Options 1 or 3 will consent to their medication and health resources use being assessed objectively over a six month period. Participants that choose Options 1 or 2 will directly provide baseline information about their health, medication use, and use of health resources via communications with researchers. Similar information will be collected directly from participants in this group after six months.

Random group allocation:

Options 1 and 2: i) Sleepwell package; ii) Empower package; iii) No package Option 3: i) Sleepwell package; ii) No package

The investigators will compare the rates of reducing and stopping sleeping pill use among the different groups over 6 months. Safety outcomes including falls and hospital visits will be measured. The investigators will also track participant access to online CBTi resources using Google Analytics.

Encouraging results from this study of direct-to-patient health promotion regarding insomnia management and sleeping pill use can be utilized repeatedly over time to reach all individuals who could benefit from the intervention, leading a transformational change in insomnia management.

ELIGIBILITY:
Inclusion Criteria:

* residents of New Brunswick, Canada
* age 65 or older
* English speaking
* community dwelling with no anticipated change of address for the next 6 months
* current user of BZRAs (3 or more bedtime doses in previous 7 days)
* long-term user of BZRA: use 3 months or longer
* BZRA indication: insomnia.

Exclusion Criteria:

* using non-BZRA sedative-hypnotics for treating insomnia or related sleep problems (e.g., trazodone, quetiapine, tricyclic antidepressant, mirtazapine, melatonin, diphenhydramine, dimenhyrdinate)
* use of alcohol or cannabis 3 or more nights a week for sleep problems
* diagnosis of other sleep disorders: sleep terrors, sleep apnea, restless legs syndrome, narcolepsy, sleepwalking
* severe anxiety disorder
* obsessive compulsive disorder
* severe cognitive impairment
* dementia
* seizure disorder
* spinal injury
* chronic psychotic disorder (e.g., schizophrenia)
* bipolar disorder
* cancer
* receiving palliative care
* living in a Long Term Care facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 594 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants discontinuing BZRA treatment within 6 months | 6 months

SECONDARY OUTCOMES:
Number of participants discontinuing BZRA treatment within 3 months | 3 months
Number of participants with BZRA dose change of 25% or more within 6 months | 6 months
  Relative change in BZRA dose between baseline and 6 months is 25% or greater.
Number of participants starting a new non-BZRA sedative-hypnotic | 6 months
  Newly started on other sedative-hypnotics

OTHER OUTCOMES:
Score on the Beliefs about Medicines Questionnaire (BMQ) | baseline, 6 months
  BMQ
Number of visits to mysleepwell.ca website | 6 months
  The count of website visits by study participants in the Sleepwell arm during 6 months
Time to fall asleep (minutes) | baseline, 6 mo.
  Sleep onset latency (SOL) measured in minutes
Time spent asleep (minutes) | baseline, 6 months
  Total sleep time (TST) measured in minutes
Sleep efficiency (%) | baseline, 6 months
  Time spent sleeping (min.) compared to total time spent in bed (min) x 100
Score on the Epworth Sleepiness Scale | baseline, 6 months
  Assessment of daytime sleepiness
Score on the Insomnia Severity Index | baseline, 6 months
Score on the Generalized anxiety disorder - 7 | baseline, 6 months
Vulnerable elderly survey, 13-item version | baseline, 6 months
  A function-based self-reported brief survey to assess risk of functional decline and death
Score on the Quality of life SF-12v2 | baseline, 6 mo.
Number of participants reporting having a fall (subjective) | baseline, 6 months
Number of participants reporting having a fall-related health visit | baseline, 6 months
Responses to the prescriber acceptability survey | 6 months
  Prescribers will be invited to respond to this end-of-study survey assessing their acceptability of the Sleepwell intervention. The development of this survey was informed by the Theoretical Framework of Acceptability

CONTACTS AND LOCATIONS:
Overall Officials: David M Gardner, PharmD, Principal Investigator — Dalhousie University
Locations (1):
- University of New Brunswick, Fredericton, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gardner DM, Turner JP, Magalhaes S, Rajda M, Murphy AL. Patient Self-Guided Interventions to Reduce Sedative Use and Improve Sleep: The YAWNS NB Randomized Clinical Trial. JAMA Psychiatry. 2024 Dec 1;81(12):1187-1197. doi: 10.1001/jamapsychiatry.2024.2731. PMID 39292452
- [Derived] Murphy AL, Turner JP, Rajda M, Magalhaes S, Allen KG, Gardner DM. A protocol for a randomized controlled trial comparing Sleepwell, EMPOWER, and treatment-as-usual for benzodiazepine receptor agonist discontinuation in older adults: the your answers when needing sleep in New Brunswick (YAWNS NB) study. Explor Res Clin Soc Pharm. 2022 Aug 3;7:100164. doi: 10.1016/j.rcsop.2022.100164. eCollection 2022 Sep. PMID 36045710